CLINICAL TRIAL: NCT01628016
Title: A Randomized, Double-blind, Placebo-Controlled Evaluation of the Efficacy of Attentional Bias Modification Training in the Treatment of Depressive Symptoms
Brief Title: The Effect of Attention Bias Modification Training on Reducing Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunan Normal University (Other)
Responsible Party: Principal Investigator, Wenhui Yang, Department of Psychology, Hunan Normal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJK011AXL002
Record Dates: First submitted 2012-06-09; First posted 2012-06-26 (Estimated); Results first posted 2019-09-19 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Depressive Symptoms
Keywords: depression; attention; training; modification
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Attentional bias modification training (Experimental): 1. Attention bias modification training (ABMT) is a modified dot probe task, in which a probe always appears in the location of neutral stimulus after the two stimuli (i.e. one is the depressive cue and the other is neutral) were simultaneously presented. In the ABMT,the probability that a probe appears in the location of neutral is 90%, and correspondingly,in the location of depressive stimuli is 10%.
  2. ABMT intervention: Participants complete 8 sessions of attention bias modification training (ABMT) during a two-week period. Each session consists of 218 trials, and the time to complete a training session is 12 minutes (4 sessions a week, roughly one session every other day with for each session).
  Interventions: Behavioral: a word dot-probe task for training procedure
- Placebo training (Placebo Comparator): Participants complete 8 sessions of placebo training(PT) during a two-week period. Placebo training is a classic dot probe task, in which a probe appears after either of the locations that the two stimuli (i.e. one is the depressive cue and the other is neutral) were presented, with the same frequencies. In the PT condition, each session also consists of 218 trials, and the time to complete a PT session is approximately 10 minutes as well.
  Interventions: Behavioral: a word dot-probe task for training procedure
- blank control (No Intervention): Participants only complete assessment at each point time.

INTERVENTIONS:
Behavioral: a word dot-probe task for training procedure — In the word dot-probe task for training procedure of attention bias modification, 90% of the targets appeared at the neutral word position and 10% at the sad word position.In the placebo condition, the targets appeared with equal probability in the sad (50%) and neutral (50%) word positions.All participants in ABM and placebo conditions received eight 12-min training sessions over a 2-week period.During each session, participants completed 216 word dot-probe trials.
  Arms: Attentional bias modification training; Placebo training

SUMMARY:
The purpose of this study is to test whether attention bias modification training is an effective neurobehavioral therapy to improve depressive symptoms.That is whether attention bias modification training is superior to placebo in reducing depressive symptoms over 1 year after training.

DETAILED DESCRIPTION:
Attentional bias has been theorized to play a critical role in the onset and maintenance of depression. Attentional bias modification training (ABMT), an experimental paradigm that uses training to induce adaptive attentional bias, was developed to test the causal model and this has therapeutic implications in depression.To test the effect of ABMT on treatment of depressive symptoms, a randomized, double-blind, placebo and blank controlled trial is conducted in college students who are experiencing mild-to-severe symptoms of depression.

ELIGIBILITY:
Inclusion Criteria:

* A score of 14 or higher on the Beck Depression Inventory-II

Exclusion criteria :

1. a current episode of MDD, bipolar disorder, schizophrenia or organic mental disorder;
2. any concurrent psychotherapy;
3. any concurrent psychotropic medication.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2011-09; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wenhui Yang, Ph.D, Principal Investigator — Department of Psychology, Hunan Normal University
Locations (1):
- Department of Psychology, Hunan Normal University, Changsha, Hunan, China

REFERENCES:
- [Derived] Yang W, Ding Z, Dai T, Peng F, Zhang JX. Attention Bias Modification training in individuals with depressive symptoms: A randomized controlled trial. J Behav Ther Exp Psychiatry. 2015 Dec;49(Pt A):101-11. doi: 10.1016/j.jbtep.2014.08.005. Epub 2014 Sep 8. PMID 25245928

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The training sessions were held in Hunan Normal University from September 14 - October 1, 2011.
Pre-assignment Details: Participants were randomly assigned to one of the three conditions by a computer-generated random assignment. Randomization was stratified by depression severity and gender.
Groups:
- Attentional Bias Modification Training: Participants complete 8 sessions of attention bias modification training (ABMT) during a two-week period. Each session consists of 218 trials, and the time to complete a training session is 12 minutes (4 sessions a week, roughly one session every other day with for each session).
  a word dot-probe task for training procedure: In the word dot-probe task for training procedure of attention bias modification, 90% of the targets appeared at the neutral word position and 10% at the sad word position.In the placebo condition, the targets appeared with equal probability
Period: Pretraining to Posttraining
Arm/Group | Attentional Bias Modification Training | Placebo Training | Blank Control
Started | 27 | 27 | 23
Completed | 27 | 27 | 23
Not Completed | 0 | 0 | 0
Period: Posttraining to 5 Follow-ups
Arm/Group | Attentional Bias Modification Training | Placebo Training | Blank Control
Started | 27 | 27 | 23
Completed | 23 | 20 | 18
Not Completed | 4 | 7 | 5

BASELINE CHARACTERISTICS:
Groups:
- Attentional Bias Modification Training: Participants complete 8 sessions of attention bias modification training (ABMT) during a two-week period. The task was a modified dot-probe task, in which 90% of the targets appeared at the neutral word position and 10% at the sad word position. Each session consists of 218 trials, and the time to complete a training session is 12 minutes (4 sessions a week, roughly one session every other day with for each session).
- Placebo Training: .Participants complete 8 sessions of placebo training(PT) during a two-week period.The placebo training procedure is a classic dot probe task in which the targets appeared with equal probability in the sad (50%) and neutral (50%) word positions.Each session consists of 218 trials, and the time to complete a PT session is approximately 12 minutes as well.The stimuli is identical to ABM condition.
- Assessment-only Control: Participants only complete assessment at each point time.
- Total: Total of all reporting groups
Arm/Group | Attentional Bias Modification Training | Placebo Training | Assessment-only Control | Total
Number analyzed (Participants) | 27 | 27 | 23 | 77
Age, Continuous [Mean (Standard Deviation); unit: years]
  age | 19.44 (1.58) | 19.52 (0.89) | 19.57 (0.73) | 19.57 (0.87)
Age, Categorical [Count of Participants; unit: Participants] — Classification of age features
  Participants
    <=18 years | 3 | 2 | 1 | 6
    Between 18 and 65 years | 24 | 25 | 22 | 71
    >=65 years | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 17 | 18 | 55
  Male | 7 | 10 | 5 | 22
Region of Enrollment [Number; unit: participants]
  China | 27 | 27 | 23 | 77

OUTCOME MEASURES:

1. Primary Outcome: Depressive Symptoms Measured by Beck Depression Inventory-II
Description: Beck Depression Inventory-II(BDI-II) contains 21 items and rates the depressive symptoms for the past two weeks. Each question provides for a response of 0 to 3. A zero response means the depressive symptom is not present; a 1 means the symptom is present, a 2 means the symptom is moderate, and a 3 means the symptom is severe. The total BDI-II score is the sum of the individual items; total BDI-II scores can range from 0 to 63. Cutoff points developed by Beck, Steer, & Brown (1997) for the total BDI-II are: 0 to 13, nondepressed; 14 to 19, mild depression; 20 to 28, moderate depression; 29 or more, severe depression.
Time Frame: From the baseline to posttraining, 2-, 4-, 8-week, 3-, 7-month follow-ups after training
Population: Some subjects dropped out of the study or could not be contacted.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Attentional Bias Modification Training: The training procedure of attention bias modification is a modified dot-probe task,in which 90% of the targets appeared at the neutral word position and 10% at the sad word position. Participants complete 8 sessions of attention bias modification training (ABMT) during a two-week period. Each session consists of 218 trials, and the time to complete a training session is 12 minutes (4 sessions a week, roughly one session every other day with for each session).
- Placebo Training: Placebo training procedure is a classic dot probe task, in which the targets appeared with equal probability in the sad (50%) and neutral (50%) word positions.Participants complete 8 sessions of placebo training(PT) during a two-week period and each session consists of 218 trials.The stimuli was identical to the ABM condition.
Arm/Group | Attentional Bias Modification Training | Placebo Training | Blank Control
Number analyzed (Participants) | 27 | 27 | 23
units on a scale
  BDI-II scores at baseline | 17.33 (3.81) | 18.04 (4.11) | 18.13 (5.18)
  BDI-II scores at posttraining | 10.96 (4.62) | 16.78 (5.09) | 18.13 (6.33)
  BDI-II scores 2-week follow-up;n=23,21,20: number analyzed (Participants) | 23 | 21 | 20
  BDI-II scores 2-week follow-up;n=23,21,20 | 9.22 (4.81) | 17.29 (6.40) | 17.00 (4.60)
  4-week follow-up;n=23,21,21: number analyzed (Participants) | 23 | 21 | 21
  4-week follow-up;n=23,21,21 | 8.26 (3.97) | 17.29 (6.40) | 17.00 (4.60)
  8-week follow-up;n=27,27,23 | 9.41 (4.56) | 17.44 (4.56) | 17.35 (5.02)
  3-momth follow-up;n=27,27,21: number analyzed (Participants) | 27 | 27 | 21
  3-momth follow-up;n=27,27,21 | 9.56 (4.56) | 14.41 (7.12) | 13.38 (5.97)
  7-month follow-up;n=23,20,18: number analyzed (Participants) | 23 | 20 | 18
  7-month follow-up;n=23,20,18 | 8.95 (4.68) | 13.20 (7.95) | 10.56 (7.35)
Statistical Analysis 1: Comparison: Attentional Bias Modification Training vs Placebo Training vs Blank Control; Test type: Other; p = .05, Mixed Models Analysis; Mean Difference (Final Values) = 3.98

2. Secondary Outcome: Anxiety and Rumination Symptoms Measured by State-Trait Anxiety Inventory-Trait(STAI-T) and Rumination Response Style（RRS）
Description: State-Trait Anxiety Inventory-Trait (STAI-T) measures the anxiety symptoms of the individuals who often feel.It consists of 20 items and each question provides for a response of 1 to 4. A 1 response means the anxiety symptom is not present; a 2 means the symptom is present but a little, a 3 means the symptom is usually present, and a 4 means the symptom lasts all the time. The total STAI-T score is the sum of the individual items; total STAI-T scores can range from 20 to 80. The higher values represent a worse outcome.
  The RRS measures ruminative responses to depressed mood. The content of the items is related to depressive cognitions and their possible causes and consequences. The scale consists of 21items and each question provides for a response of 1 to 4. The total RRS scores can range from 21 to 84. The higher values represent a worse outcome.
Time Frame: From baseline to post-training, 2-, 4-, 8-week, 3- , 7-month follow-ups after training
Population: Some subjects dropped out of the study or could not be contacted.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Attentional Bias Modification Training: Participants complete 8 sessions of attention bias modification training (ABMT) during a two-week period. Each session consists of 218 trials, and the time to complete a training session is 12 minutes (4 sessions a week, roughly one session every other day with for each session).
- Placebo Training: Participants complete 8 sessions of placebo training(PT) during a two-week period.
Arm/Group | Attentional Bias Modification Training | Placebo Training | Blank Control
Number analyzed (Participants) | 27 | 27 | 23
units on a scale
  STAI-T score at postraining;n=27,27,23 | 44.52 (4.56) | 50.81 (5.20) | 51.35 (5.46)
  STAI-T score at 2-week follow-up;n=23,21,20: number analyzed (Participants) | 23 | 21 | 20
  STAI-T score at 2-week follow-up;n=23,21,20 | 43.82 (4.21) | 50.23 (7.48) | 50.30 (5.51)
  STAI-T score at 4-week follow-up;n=23,21,21: number analyzed (Participants) | 23 | 21 | 21
  STAI-T score at 4-week follow-up;n=23,21,21 | 44.39 (4.28) | 50.05 (6.82) | 50.05 (5.63)
  STAI-T score at 8-week follow-up;n=27,27,23 | 44.15 (4.67) | 49.19 (6.14) | 50.13 (5.74)
  STAI-T score at 3-month follow-up;n=27,27,21: number analyzed (Participants) | 27 | 27 | 21
  STAI-T score at 3-month follow-up;n=27,27,21 | 44.74 (5.20) | 47.41 (7.42) | 46.82 (7.86)
  STAI-T score at 7-month follow-up;n=23,20,18: number analyzed (Participants) | 23 | 20 | 18
  STAI-T score at 7-month follow-up;n=23,20,18 | 47.87 (5.31) | 48.25 (6.38) | 45.94 (6.79)
  RRS score at postraining;n=27,27,23 | 41.40 (5.44) | 45.44 (8.08) | 46.78 (6.27)
  RRS score at 2-week follow-up;n=23,21,20: number analyzed (Participants) | 23 | 21 | 20
  RRS score at 2-week follow-up;n=23,21,20 | 41.22 (4.45) | 45.52 (7.78) | 46.50 (6.61)
  RRS score at 4-week follow-up;n=23,21,21: number analyzed (Participants) | 23 | 21 | 21
  RRS score at 4-week follow-up;n=23,21,21 | 38.91 (4.16) | 45.14 (7.47) | 46.33 (6.26)
  RRS score at 8-week follow-up;n=27,27,23 | 39.07 (5.17) | 44.29 (8.09) | 45.57 (6.51)
  RRS score at 3-month follow-up;n=27,27,21: number analyzed (Participants) | 27 | 27 | 21
  RRS score at 3-month follow-up;n=27,27,21 | 42.96 (6.08) | 44.15 (8.11) | 45.52 (7.37)
  RRS score at 7-month follow-up;n=23,20,18: number analyzed (Participants) | 23 | 20 | 18
  RRS score at 7-month follow-up;n=23,20,18 | 43.43 (6.75) | 46.75 (8.87) | 44.22 (7.92)

ADVERSE EVENTS:
Time Frame: 7-month
Arm/Group | Attentional Bias Modification Training | Placebo Training | Blank Control
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/23
Other Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No